CLINICAL TRIAL: NCT04740398
Title: A Phase Ia/Ib, Open-Label, Multi-center, First in Human and Expansion Study to Assess the Safety, Tolerance, and Pharmacokinetics of the Novel Antitumor Agent CBP-1008 in Patients With Advanced Solid Tumors
Brief Title: A Study of CBP-1008 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Coherent Biopharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP-1008-01
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ia stage - CBP-1008 Dose escalation/ Ib stage - CBP-1008 monotherapy (Experimental): Ia:Patients will receive CBP-1008 IV infusion every 2 weeks until disease progression, intolerability, informed consent withdraw, or other reasons leading to treatment discontinue.
  Ib:Patients will receive CBP-1008 RP2D IV infusion every two weeks until disease progression, intolerability, informed consent withdraw, or other reasons leading to treatment discontinue.
  Interventions: Drug: CBP-1008

INTERVENTIONS:
Drug: CBP-1008 — CBP-1008 for injection; IV infusion; Infusion for 90 minutes

SUMMARY:
The primary objective of this phase I study is to evaluate the safety and potential efficacy and to determine the recommended phase 2 dose (RP2D) of CBP-1008, a bi-specific ligand conjugated drugs in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This phase Ia/Ib, open-label, multicenter study has two stages. The Ia stage is a dose-escalation study that will focus on safety, tolerability, pharmacokinetics, MTD and RP2D. Patients with advanced solid tumor who failed from previous standard treatment or without standard therapy exists will be enrolled in the phase Ia study. DLT observation period is 28 days.

Patients in phase Ib part will be recruited into certain tumor cohorts and receive RP2D CBP-1008 iv infusion every two weeks. Primary efficacy of ORR, DCR, PFS, etc., will be evaluated. The correlation between tumor response and the receptors will be explored. Safety information will be collected in phase Ib stage.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged 18-70 years (including the boundaries) when signed informed consent form (ICF)
* Has a life expectancy of ≥ 3 months
* Phase Ia: patients with advanced malignant solid tumor who:
* have progressed on or are intolerant to standard therapy, or
* no standard therapy exists
* Phase Ib disease specific Cohorts:
* Cohort 1: Platinum-resistant advanced high-grade serous ovarian cancer, fallopian tube cancer or primary peritoneal cancer.Platinum resistance was defined as progression or recurrence within 6 months after the last dose of platinum. Patients with primary platinum refractory disease are excluded
* Cohort 2: Metastatic triple-negative breast cancer
* Based on most recently analyzed biopsy or other pathological specimens, TNBC was confirmed histologically or cytologically
* Patients have received at least 2 previous systemic chemotherapy regimens for local advanced/metastasis disease. If the patients in the early phase develop into unresectable locally advanced or metastatic disease within 12 months after adjuvant or neoadjuvant chemotherapy, the regimens will be regarded as one of the previous systemic chemotherapy regimens
* Cohort 3: Patients with other advanced solid tumor types who failed from standard therapy or no standard therapy exists or intolerant to the existing treatment, such as: Esophageal squamous cell carcinoma, Non-triple-negative breast cancer, head and neck squamous cell carcinoma, lung squamous cell carcinoma, gastric adenocarcinoma, colon cancer, cervical cancer, endometrial cancer, and so on
* Cohort 4: Other types of ovarian cancer that are resistant to platinum (clear cell carcinoma and/or low-grade serous carcinoma, etc.)
* Has an Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1
* At least 1 measurable tumor lesion according to RECIST v1.1
* Archived tumor tissue samples available or fresh tumor biopsy samples available
* FOLR1 and/or TRPV6 receptor expression tested positive by the central laboratory
* The time window from the last administration of previous anti-tumor therapy to the first administration of CBP-1008 in this study was at least 28 days. No other trial drugs or experimental instruments was used or other clinical trials were conducted within 28 days before the start of trial drugs
* According to the NCI-CTCAE 4.03 version, the acute toxicity of any previous treatment, surgery or radiotherapy must have been alleviated to grade 0 or 1
* Adequate hematologic status (without receiving blood transfusion and growth factor support within 2 weeks before enrollment), defined as:
* Absolute neutrophil count (ANC) ≥ 1.5× 109/L
* Platelet count ≥ 90 × 109/L
* Hemoglobin (Hb) ≥ 95 g/L
* Adequate hepatic function, defined as:
* Serum total bilirubin (TBIL) ≤ 1.5× ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN if no demonstrable liver metastases (ALT and AST ≤ 3.0× ULN in the presence of liver metastases)
* Adequate renal function, defined as:
* Serum creatinine < upper limit of laboratory normal reference range, or creatinine clearance ≥50 mL/min/1.73㎡ (The calculation formula is shown in Appendix 11)
* Coagulation: International Normalized Ratio (INR) ≤ 1.5× ULN and activated partial thromboplastin time (APTT) ≤ 1.5× ULN (except patients who are receiving therapeutic anticoagulation, whose INR should be within the therapeutic range)
* Appropriate serum calcium concentration: Refer to serum albumin-corrected calcium concentration ≥ 1 × lower limit of normal (ULN) and ≤ 2.9 mmol/L (11.5 mg/dL) if the subjects had hypocalcemia and hypoproteinemia
* Adequate cardiac function, defined as:
* Left ventricular eject fraction (LVEF) ≥ 50% or lower limit of normal reference range in hospital
* QTc-F≤ 450 ms

Exclusion Criteria:

* History of allergic reactions to any component of the CBP-1008
* Concurrent malignancy(ies) within 3 years prior to screening other than adequately treated cervical carcinoma-in-situ, skin cancer of basal cell or squamous cell carcinoma, local prostate cancer after radical operation, ductal carcinoma in situ after radical operation
* History of epilepsy
* Active or symptomatic central nervous system metastasis and / or cancerous meningitis with the exception of, asymptomatic or stable brain metastases
* History of congestive heart failure of the New York Heart Association Functional Classification III/IV, unstable angina pectoris, persistent atrial fibrillation, ventricular arrhythmia or conduction block; with risk factors for, or are receiving medications known to prolong QT interval, refractory hypertension (except hypertension patients whose blood pressure is controlled below 140 / 90mmHg by drugs)
* Significant surgical interventions within 21 days prior to the first dose of CBP-1008 or with ongoing post-operative complications
* Radiotherapy administrated within 21 days prior to the first dose of CBP-1008
* Interstitial lung disease, non-infectious pneumonia or a history of poorly controlled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc
* Active infections requiring systemic treatment, active viral hepatitis or active tuberculosis
* Pericardial effusion with important clinical significance
* Clinically uncontrolled pleural effusion or ascites requiring drainage within 1 month before administration

  •≥level 2 Peripheral neuropathy, according to NCI CTCAE 4.03 criteria
* For subjects with lung squamous cell carcinoma, there was hemoptysis within 28 days prior to the first dose of CBP-1008 (hemoptysis volume ≥ 2.5ml each time)
* A history of gastrointestinal perforation and / or complete intestinal obstructio within 6 months prior to the first dose of CBP-1008
* There is higher risk of bleeding or fistula caused by the adjacent organs of esophageal lesions (large artery or trachea) invaded by the tumor. Subjects after endotracheal stent implantation
* Foods or drugs known as potent or moderate CYP3A inhibitors or potent CYP3A inducers which has been used 10 days before the first dose or is expected to use
* Female subject who are pregnant or breastfeeding or considering pregnancy
* Any medical situation assessed by the researcher may increase the patient's safety risk, limit study compliance or interfere with study evaluation
* Alcoholism within 3 months prior to the first dose of CBP-1008
* Known drug abuse within 6 months before signing ICF
* Human immunodeficiency virus infection (HIV-1/2 antibody positive), active hepatitis B virus (HBV) infection，hepatitis C virus (HCV) infection (HCV antibody positive) or syphilis infection. Active hepatitis B was defined as HBV DNA ≥ upper limit of laboratory normal reference range
* Other situations considered unsuitable for inclusion by the researcher

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | up to 12 months
  Assessed by number of patients with AE, Treatment-Emergent Adverse Event (TEAE), serious adverse event (SAE), and discontinuation of study drug due to AE.
To determine the maximum tolerated dose (MTD) | Up to 28 days after the first dose of CBP-1008
  Dose limiting toxicity (DLT) will be assessed by NCI CTCAE v4.03. MTD is defined as the previous dose level at which 2 out of 3 participants or 2 out of 6 participants experienced DLT.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of CBP-1008 | up to 12 months
  Maximum serum concentration (Cmax) of CBP-1008 will be investigated.
Time to maximum serum concentration (Tmax) of CBP-1008 | up to 12 months
  Tmax of CBP-1008 will be investigated.
Elimination half-life (T1/2) of CBP-1008 | up to 12 months
  T1/2 of CBP-1008 will be investigated.
AUC0-t of CBP-1008 | up to 12 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
Clearance (CL) in the serum of CBP-1008 per unit of time | up to 12 months
  CL in the serum of CBP-1008 per unit of time will be investigated.
6. The percentage of participants with anti-drug antibody (ADA) positive after dosing CBP-1008 | up to 12 months
  Incidence and titer of ADA against CBP-1008 will be evaluated.
Recommended Phase II Dose (RP2D) | up to 12 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) based on safety, tolerability, efficacy, PK data collected during the dose escalation study of CBP-1008.
Objective Response Rate (ORR) | up to 12 months
  ORR was defined as the percentage of participants, who had a CR or PR. The percentage of participants who experienced a confirmed CR or PR is evaluated by investigator according to RECIST 1.1.
Duration of Response (DOR) | up to 12 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first. The DOR is evaluated by investigator according to RECIST 1.1.
Clinical benefit rate (CBR) | up to 12 months
  CBR was defined as the percentage of participants, who had a CR, PR or SD. The percentage of participants who experienced a confirmed CR, PR or SD is evaluated by investigator according to RECIST 1.1.
Progression-free survival rate (PFS) | up to 12 months
  The PFS is defined as the time from the participant's first dose of CBP-1008 to the first date of either disease progression or death, which will be evaluated by investigator according to RECIST 1.1.
Overall survival rate (OS) | up to 12 months
  12 months OS will be evaluated by investigator according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No